CLINICAL TRIAL: NCT00793546
Title: A Phase 2, Randomized, Open-Label Study Of Bosutinib Administered In Combination With Exemestane Versus Exemestane Alone As Second Line Therapy In Postmenopausal Women With Locally Advanced Or Metastatic ER+/PgR+/ErbB2- Breast Cancer
Brief Title: Study Evaluating Bosutinib-Exemestane Combination Vs Exemestane Alone in Post Menopausal Women With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3160A6-2206; B1871009
Record Dates: First submitted 2008-10-29; First posted 2008-11-19 (Estimated); Results first posted 2012-11-05 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-10

CONDITIONS: Advanced Breast Cancer
Keywords: Bosutinib; Exemestane; postmenopausal; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — bosutinib; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): combination of bosutinib and exemestane
  Interventions: Drug: Bosutinib; Drug: exemestane
- 2 (Active Comparator): exemestane
  Interventions: Drug: Exemestane

INTERVENTIONS:
Drug: Bosutinib — 300 mg =(3x100mg) tablets once daily during the active phase of treatment until disease progression, unacceptable toxicity or withdrawal of consent occurs
  Arms: 1
Drug: exemestane — 25 mg tablet once daily
  Arms: 1
Drug: Exemestane — 25 mg - 1 tablet per day- once daily daily during the active phase of treatment until disease progression, unacceptable toxicity or withdrawal of consent occurs
  Arms: 2

SUMMARY:
This is a phase 2, open-label, multicenter, 2-arm study of bosutinib administered in combination with exemestane versus exemestane alone. This is a 2-part study consisting of a safety lead-in phase and randomized phase 2 portion. Subjects in part 1 will receive bosutinib and exemestane daily, and will be closely monitored for 28 days. If no safety concerns arise, then future eligible subjects will be randomly assigned to the main phase of the study. They will either receive bosutinib daily combined with daily exemestane, or daily exemestane alone for a specified period of time. Subjects will be followed up for survival after treatment discontinuation.

DETAILED DESCRIPTION:
This study was terminated on 19 Apr 2010 due to unfavorable risk benefit ratio which did not support continuation in part 2 of the study. Even if the safety profile of the combination of Bosutinib and Exemestane was acceptable 25% of subjects had treatment related liver events including 14% of severe liver events.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18 years or older.
* Confirmed pathologic diagnosis of breast cancer.
* Locally advanced, metastatic, or locoregional recurrent breast cancer not amenable to curative treatment with surgery or radiotherapy.
* Surgically sterile or postmenopausal woman.
* Documented ER+ and/or PgR+ and erbB2- tumor.
* Progression of locally advanced or metastatic disease during treatment with a nonsteroidal AI or tamoxifen, or progression during treatment with (or within 6 months of discontinuation of) an adjuvant nonsteroidal AI.

Exclusion Criteria:

* Prior exemestane, prior bosutinib, or any other prior anti-Src therapy.
* More than 1 prior endocrine treatment for locally advanced or MBC.
* More than 1 prior cytotoxic chemotherapy regimen in metastatic setting.
* Bone or skin as the only site of disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (9):
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Joliet, Illinois
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Seattle, Washington
- Pfizer Investigational Site, South Brisbane, Queensland, Australia
- Belgium (4):
  - Pfizer Investigational Site, Brussels, Brussels Capital
  - Pfizer Investigational Site, Leuven, Leuven
  - Pfizer Investigational Site, Liège, Liege
  - Pfizer Investigational Site, Wilrijk
- Pfizer Investigational Site, Kelowna, British Columbia, Canada
- Pfizer Investigational Site, Beijing, China
- Pfizer Investigational Site, Hong Kong, Hong Kong
- Pfizer Investigational Site, Budapest, Hungary
- India (2):
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Pune, Maharashtra
- Pfizer Investigational Site, Olsztyn, Poland
- Pfizer Investigational Site, Lynnwood, Gauteng, South Africa
- Spain (3):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Valencia, Valencia
- Pfizer Investigational Site

REFERENCES:
- [Derived] Moy B, Neven P, Lebrun F, Bellet M, Xu B, Sarosiek T, Chow L, Goss P, Zacharchuk C, Leip E, Turnbull K, Bardy-Bouxin N, Duvillie L, Lang I. Bosutinib in combination with the aromatase inhibitor exemestane: a phase II trial in postmenopausal women with previously treated locally advanced or metastatic hormone receptor-positive/HER2-negative breast cancer. Oncologist. 2014 Apr;19(4):346-7. doi: 10.1634/theoncologist.2014-0022. Epub 2014 Mar 27. PMID 24674873
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3160A6-2206&StudyName=Study%20Evaluating%20Bosutinib-Exemestane%20Combination%20Vs%20Exemestane%20Alone%20in%20Post%20Menopausal%20Women%20With%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was pre-maturely terminated after part 1 (safety lead-in phase) of the study and hence, the planned treatments of part 2, bosutinib + exemestane (part 2) and exemestane (part 2), were not administered.
Groups:
- Bosutinib 400 mg + Exemestane 25 mg (Part 1): Four bosutinib 100 milligram (mg) tablets (equivalent to 400 mg bosutinib) orally along with exemestane 25 mg tablet orally once daily up to 6 months or until disease progression, unacceptable toxicity, withdrawal of consent.
- Bosutinib 300 mg + Exemestane 25 mg (Part 1): Three bosutinib 100 mg tablets (equivalent to 300 mg bosutinib) orally along with exemestane 25 mg tablet orally once daily up to 6 months or until disease progression, unacceptable toxicity, withdrawal of consent.
Period: Overall Study
Arm/Group | Bosutinib 400 mg + Exemestane 25 mg (Part 1) | Bosutinib 300 mg + Exemestane 25 mg (Part 1)
Started | 14 | 28
Completed | 0 | 0
Not Completed | 14 | 28
Not completed — Death | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Study Terminated by Sponsor | 8 | 27
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bosutinib 400 mg + Exemestane 25 mg (Part 1) | Bosutinib 300 mg + Exemestane 25 mg (Part 1) | Total
Number analyzed (Participants) | 14 | 28 | 42
Age Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.16) | 58.2 (10.02) | 60.2 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 28 | 42
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Based on Independent Radiologist
Description: Time in weeks from randomization to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of randomization plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Part 2 Baseline, every 8 weeks up to 2 to 6 weeks after last dose
Population: Data were not analyzed because the study was prematurely terminated due to unfavorable risk benefit ratio of the study treatment.
Groups:
- Bosutinib 300 mg + Exemestane 25 mg (Part 2): Three bosutinib 100 mg tablets (equivalent to 300 mg bosutinib) orally along with exemestane 25 mg tablet orally once daily up to 6 months or until disease progression, unacceptable toxicity, withdrawal of consent.
- Exemestane 25 mg (Part 2): Exemestane 25 mg tablet orally once daily up to 6 months or until disease progression, unacceptible toxicity or withdrawal of consent.
Arm/Group | Bosutinib 300 mg + Exemestane 25 mg (Part 2) | Exemestane 25 mg (Part 2)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) And Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 28 days after the last dose
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib 400 mg + Exemestane 25 mg (Part 1) | Bosutinib 300 mg + Exemestane 25 mg (Part 1)
Number analyzed (Participants) | 14 | 28
percentage of participants
  AEs | 100 | 96.4
  SAEs | 28.6 | 17.9

3. Secondary Outcome: Progression Free Survival (PFS) Based on Investigator
Description: as for outcome 1
Time Frame: Part 2 Baseline, every 8 weeks up to 2 to 6 weeks after last dose
Population: as for outcome 1
Arm/Group | Bosutinib 300 mg + Exemestane 25 mg (Part 2) | Exemestane 25 mg (Part 2)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as greater than or equal to >=30 percent (%) decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study >=4 weeks after initial documentation of response.
Time Frame: Part 2 Baseline, every 8 weeks up to 2 to 6 weeks after last dose
Population: as for outcome 1
Arm/Group | Bosutinib 300 mg + Exemestane 25 mg (Part 2) | Exemestane 25 mg (Part 2)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Time in weeks from randomization to date of death due to any cause. OS was calculated as (the death date minus the date of randomization plus 1) divided by 7. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Part 2 Baseline until death or up to 24 months
Population: as for outcome 1
Arm/Group | Bosutinib 300 mg + Exemestane 25 mg (Part 2) | Exemestane 25 mg (Part 2)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Part 2 Baseline, every 8 weeks up to 2 to 6 weeks after last dose
Population: as for outcome 1
Arm/Group | Bosutinib 300 mg + Exemestane 25 mg (Part 2) | Exemestane 25 mg (Part 2)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B)
Description: FACT-B is used for assessment of health-related quality of life (QoL) in participants with breast cancer. It consists of 36 items, summarized to 5 subscales: physical (7 items), functional (7 items), social/family (7 items); all 3 ranged from 0 to 28, emotional (6 items) ranging from 0 to 24, and additional concerns on breast cancer subscale (9 items) ranging from 0 to 36; high subscale score represents a better QoL. All single-item measures ranges from 0='Not at all' to 4='Very much'. Total possible score ranged from 0 to 144. High scale score represents a better QoL.
Time Frame: Part 2 Baseline, Week 12, 2 to 6 weeks after last dose
Population: as for outcome 1
Arm/Group | Bosutinib 300 mg + Exemestane 25 mg (Part 2) | Exemestane 25 mg (Part 2)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Euro Quality of Life (EQ-5D)- Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Part 2 Baseline, Week 12, 2 to 6 weeks after last dose
Population: as for outcome 1
Arm/Group | Bosutinib 300 mg + Exemestane 25 mg (Part 2) | Exemestane 25 mg (Part 2)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Euro Quality of Life (EQ-5D)- Visual Analog Scale (VAS)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 millimeter (mm) = worst imaginable health state to 100 mm =best imaginable health state; higher scores indicate a better health state.
Time Frame: Part 2 Baseline, Week 12, 2 to 6 weeks after last dose
Population: as for outcome 1
Arm/Group | Bosutinib 300 mg + Exemestane 25 mg (Part 2) | Exemestane 25 mg (Part 2)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 hour (pre-dose) on Day 1, 1, 2, 3, 4, 6, 8, 24 hours post-dose on Day 29
Population: as for outcome 1
Arm/Group | Bosutinib 300 mg + Exemestane 25 mg (Part 2) | Exemestane 25 mg (Part 2)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 hour (pre-dose) on Day 1, 1, 2, 3, 4, 6, 8, 24 hours post-dose on Day 29
Population: as for outcome 1
Arm/Group | Bosutinib 300 mg + Exemestane 25 mg (Part 2) | Exemestane 25 mg (Part 2)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-24)]
Description: AUC (0-24)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-24).
Time Frame: 0 hour (pre-dose) on Day 1, 1, 2, 3, 4, 6, 8, 24 hours post-dose on Day 29
Population: as for outcome 1
Arm/Group | Bosutinib 300 mg + Exemestane 25 mg (Part 2) | Exemestane 25 mg (Part 2)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Bosutinib 400 mg + Exemestane 25 mg (Part 1) | Bosutinib 300 mg + Exemestane 25 mg (Part 1)
Serious Adverse Events (participants affected / at risk) | 4/14 | 5/28
Other Adverse Events (participants affected / at risk) | 14/14 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib 400 mg + Exemestane 25 mg (Part 1) (N=14) | Bosutinib 300 mg + Exemestane 25 mg (Part 1) (N=28)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
General physical health deterioration (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib 400 mg + Exemestane 25 mg (Part 1) (N=14) | Bosutinib 300 mg + Exemestane 25 mg (Part 1) (N=28)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 9
Diarrhoea (Gastrointestinal disorders) | 12 | 15
Dyspepsia (Gastrointestinal disorders) | 1 | 5
Nausea (Gastrointestinal disorders) | 11 | 15
Vomiting (Gastrointestinal disorders) | 8 | 12
Asthenia (General disorders) | 3 | 3
Fatigue (General disorders) | 4 | 6
Oedema peripheral (General disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 4 | 7
Aspartate aminotransferase increased (Investigations) | 3 | 4
Blood creatinine increased (Investigations) | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Dizziness (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 3 | 4
Insomnia (Psychiatric disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 4
Hot flush (Vascular disorders) | 0 | 4

LIMITATIONS AND CAVEATS:
Results are not provided because the study was terminated prior to part 2 due to unfavorable risk benefit ratio of the study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.